CLINICAL TRIAL: NCT00252408
Title: Danish Osteoporosis Prevention Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Karen Elise Jensen Foundation (Other); Novo Nordisk A/S (Industry); LEO Pharma (Industry); Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1990/1821; DOPS
Record Dates: First submitted 2005-11-10; First posted 2005-11-11 (Estimated); Last update posted 2009-09-04 (Estimated); Status verified 2009-09

CONDITIONS: Osteoporosis
Keywords: Fracture; Osteoporosis; Bone mineral density; Hormone replacement therapy; Estrogen; Breast cancer
MeSH Terms: conditions — Osteoporosis; Fractures, Bone; Breast Neoplasms | interventions — Hormone Replacement Therapy

INTERVENTIONS:
Drug: Hormone replacement therapy

SUMMARY:
Hypothesis: Use of hormone replacement therapy (HRT) decreases the incidence of fractures in early postmenopausal women.

The project was initiated in 1990, and the inclusion ended in 1993. A total of 2,016 early postmenopausal women were divided into two groups: The first group accepted randomisation to HRT or not, and the second group was allowed to choose HRT or not.

The study was not blinded. Main measurements were fracture risk over 20 years, changes in bone mineral density over 20 years, and side effects, mainly breast cancer.

DETAILED DESCRIPTION:
Aim: To study the ability of hormone replacement early after menopause on risk of fractures and changes in bone mineral density, and side effects.

The project was designed as a comprehensive cohort trial. One group accepted randomisation, and was randomised to hormone replacement therapy (HRT) or not (no placebo used).

502 were randomised to HRT, and 504 were randomised to no HRT) One group was allowed to choose HRT or not. A total of 221 chose HRT, and 789 chose no HRT.

First line HRT was oral sequential oestradiol/norethisterone in women with intact uterus and oral continuous oestradiol in hysterectomised women.

The study was initiated in 1990, and inclusion ended in 1993.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 45-58 years with an intact uterus
* Three to 24 month past last menstrual bleeding
* Hysterectomised women aged 45-52 years and having elevated FSH

Exclusion Criteria:

* Metaboliv bone disease including osteoporosis defined as non-traumatic vertebral fractures on X-ray
* Current estrogen use or estrogen use within the past three month
* Current or past treatment with glucocorticoids for more than 6 month
* Current or past malignancy
* Newly diagnosed or uncontrolled chronic disease
* Alcohol or drug addiction

Ages: 45 Years to 58 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2000
Dates: Start 1990-10; Study Completion 2003-12

PRIMARY OUTCOMES:
Fracture
Bone mineral density

SECONDARY OUTCOMES:
Breast cancer
Menopausal symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Leif Mosekilde, Professor MD DrMedSc, Study Chair — department of Endocrinology and Metabolism C, Aarhus University Hospital, Denmark; Jens Erik Beck Jensen, MD PhD, Study Director — The Osteoporosis Clinic, Hvidovre Hospital, Copenhagen; Peder Charles, MD DrMedSc, Study Director — Department of Endocrinology and Metabolism C, Aarhus University Hospital, Denmark; Stig Pors Nielsen, MD DrMedSc, Study Director — Department of Clinical Physiology and Nuclear Medicine, Hillerød Hospital, Hillerød, Denmark; Henning Beck Nielsen, MD DrMedSc, Study Director — Odense University Hospital; Kim Brixen, MD PhD, Study Director — Odense University Hospital; Ole Helmer Sørensen, MD DrMedSc, Study Director — The Osteoporosis Clinic, Hvidovre Hospital, Copenhagen, Denmark
Locations (1):
- The Osteoporosis Clinic, Aarhus Sygehus, Aarhus, Denmark

REFERENCES:
- [Result] Mosekilde L, Beck-Nielsen H, Sorensen OH, Nielsen SP, Charles P, Vestergaard P, Hermann AP, Gram J, Hansen TB, Abrahamsen B, Ebbesen EN, Stilgren L, Jensen LB, Brot C, Hansen B, Tofteng CL, Eiken P, Kolthoff N. Hormonal replacement therapy reduces forearm fracture incidence in recent postmenopausal women - results of the Danish Osteoporosis Prevention Study. Maturitas. 2000 Oct 31;36(3):181-93. doi: 10.1016/s0378-5122(00)00158-4. PMID 11063900
- [Derived] Torekov SS, Harslof T, Rejnmark L, Eiken P, Jensen JB, Herman AP, Hansen T, Pedersen O, Holst JJ, Langdahl BL. A functional amino acid substitution in the glucose-dependent insulinotropic polypeptide receptor (GIPR) gene is associated with lower bone mineral density and increased fracture risk. J Clin Endocrinol Metab. 2014 Apr;99(4):E729-33. doi: 10.1210/jc.2013-3766. Epub 2014 Jan 21. PMID 24446656
- [Derived] Schierbeck LL, Rejnmark L, Tofteng CL, Stilgren L, Eiken P, Mosekilde L, Kober L, Jensen JE. Effect of hormone replacement therapy on cardiovascular events in recently postmenopausal women: randomised trial. BMJ. 2012 Oct 9;345:e6409. doi: 10.1136/bmj.e6409. PMID 23048011